CLINICAL TRIAL: NCT05962749
Title: The Relationship of Forward and Backward Walking with Selective Motor Control, Trunk Control and Balance in Children with Cerebral Palsy
Brief Title: The Relationship of Forward and Backward Walking with SMC, Trunk Control and Balance in Children with Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ebru Keklikci, Research Assistant, Alanya Alaaddin Keykubat University
Other Study IDs: 2023-743
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy; Balance; Gait Disorders in Children
Keywords: Cerebral Palsy; Backward Walking; Selective Motor Control; Trunk Control; Balance
MeSH Terms: conditions — Cerebral Palsy | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children With Cerebral Palsy
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — 3 meter backward walk test (3MBWT), 10 meter walk test (10MWT), Selective Control Assessment of the Lower Extremities (SCALE), Trunk Control Measurement Scale (TCMS), Pediatric Balance Scale (PBS), Functional Independence Measure for Children (WeeFIM), Modified Ashworth Scale (MAS)

SUMMARY:
Children aged between 6-18 years old, diagnosed with cerebral palsy and meeting the inclusion criteria, will be included in this study. All children and their parents who agree to participate in the study will be informed about the study and will be required to sign an "Informed Consent Form" indicating their voluntary participation.

To evaluate gait, the 3-Meter Backward Walking Test (3MBWT) and the 10-Meter Walk Test (10MWT) will be performed on a flat. The Selective Control Assessment of the Lower Extremity (SCALE) will be used to assess selective motor control in the lower extremity (hip, knee, ankle, subtalar, and toe joints). To evaluate trunk control, the Trunk Control Measurement Scale (TCMS) will be applied in a sitting position. For balance assessment, the Pediatric Balance Scale will be used to reflect activities of daily living. To assess functional independence, the Pediatric Functional Independence Measure (WeeFIM) will be applied. The Modified Ashworth Scale (MAS) will be used to evaluate muscle spasticity.

DETAILED DESCRIPTION:
Children aged between 6-18 years old, diagnosed with cerebral palsy and meeting the inclusion criteria, will be included in this study. The study will be conducted at the Özel Özgün Kardelen Special Education and Rehabilitation Center, affiliated with the Ministry of National Education in Antalya. All children and their parents who agree to participate in the study will be informed about the study and will be required to sign an "Informed Consent Form" indicating their voluntary participation.

To evaluate gait, the 3-Meter Backward Walking Test (3MBWT) and the 10-Meter Walk Test (10MWT) will be performed on a flat, obstacle-free track measuring 3 meters and 10 meters in length. The Selective Control Assessment of the Lower Extremity (SCALE) will be used to assess selective motor control in the lower extremity (hip, knee, ankle, subtalar, and toe joints). To evaluate trunk control, the Trunk Control Measurement Scale (TCMS) will be applied in a sitting position.

For balance assessment, the Pediatric Balance Scale, consisting of 14 items with increasing difficulty from a sitting position to standing on one leg, will be used to reflect activities of daily living. To assess functional independence, the Pediatric Functional Independence Measure (WeeFIM), which includes 6 sections and 18 items, will be applied. The Modified Ashworth Scale (MAS) will be used to evaluate muscle spasticity.

Each child will be assessed only once. Statistical analyses for the study will be conducted using the Statistical Package for Social Sciences (SPSS) Version 21.0 (SPSS Inc., Chicago, IL, USA). Data distribution will be examined using the Shapiro-Wilk Test. Variables with normal distribution will be presented as mean ± standard deviation, while non-normally distributed variables will be presented as median (IQR). Categorical variables will be expressed as frequency and percentage (%). The correlation between the assessment results in the cases will be determined based on the normality of the distribution. The statistical error level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with cerebral palsy by a specialist physician
* Gross Motor Function Classification System (GMFCS) level I or II
* Children with lower extremity muscles level ≤ 2 according to the Modified Ashworth Scale (MAS)
* Ability to follow verbal commands
* Modified Ashworth Scale (MAS) Level ≤2
* Complete passive range of motion in the ankle and knee joints
* Agree to participate in the study (with parent and child consent)

Exclusion Criteria:

* Having had Botox (Botulinum toxin) or a surgical operation in the last 6 months
* Having contractures in the ankle and knee joints that affect walking

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who apply for rehabilitation in Special Education and Rehabilitation Centers affiliated to the Ministry of National Education in the city of Antalya will be included in the study.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
3 meter backward walk test (3MBWT) | First day
  The 3-Meter Backward Walk Test (3MBWT) measures the time it takes for a person to walk 3 meters backward. This test assesses balance, coordination, and leg strength, making it especially useful for individuals at risk of falling or those with neurological issues. During the test, the participant is timed while walking backward over a flat 3-meter distance. Completing the distance quickly and safely indicates good balance and backward walking ability, while taking longer may suggest potential issues with balance or motor control. This simple yet effective test is used in clinical settings to evaluate functional mobility and monitor progress over time.
10 meter walk test (10MWT) | First day
  The 10-Meter Walk Test (10MWT) measures the time it takes for a person to walk a distance of 10 meters at their comfortable walking pace. This test is widely used to assess walking speed, gait, and functional mobility, and it can be particularly beneficial for individuals with mobility impairments, including those with neurological conditions or musculoskeletal issues. During the test, the participant is timed while walking the 10-meter distance, with the time recorded starting when the participant's foot crosses the starting line and stopping when they cross the finish line. A shorter completion time indicates better walking speed and mobility, while longer times may suggest difficulties in gait or increased risk of falls. The 10MWT is a straightforward and effective tool used in clinical settings to evaluate functional mobility and track changes over time.

SECONDARY OUTCOMES:
Selective Control Assessment of the Lower Extremities (SCALE) | First day
  While applying the Selective Control Assessment of the Lower Extremities (SCALE), the child is asked to perform specific isolated movement patterns at the hip, knee, ankle, subtalar, and toe joints. The clinician scores the selective motor control of each joint based on the child's ability to perform isolated movements. The child receives 2 points if they can move the tested joint in isolation, 1 point if mirror movements occur, indicating impaired selectivity in the untested joint, and 0 points if no movement occurs in the tested joint or if mass-synergy patterns are present. A low score on the SCALE indicates poor selective motor control in the lower extremities.
Trunk Control Measurement Scale (TCMS) | First day
  The Trunk Control Measurement Scale (TCMS) is a clinical tool used to assess trunk control and sitting balance during functional activities. It consists of 15 items that evaluate a person's ability to maintain trunk stability in different positions and movements, making it particularly useful for individuals with neurological conditions, such as stroke or cerebral palsy. During the test, the participant is asked to perform various tasks, such as reaching, turning, and maintaining balance while sitting. Each item is scored, contributing to a total score, with higher scores indicating better trunk control and balance.
Pediatric Balance Scale (PBS) | First day
  The 'Pediatric Balance Scale (PBS)' has 14 items of increasing difficulty to test functional skills related to activities of daily living from sitting to standing on one leg. Each item is scored on a five-point ordinal scale ranging from 0 to 4 points, with a maximum score level of 56. Higher scores indicate better balance.
Functional Independence Measure for Children (WeeFIM) | First day
  The 'Functional Independence Measure for Children (WeeFIM)' has 6 sections, namely sphincter control, self-care, communication, locomotion, social cognition and transfers. There are a total of 18 items in these sections and each item is scored from 1 to 7. Scoring is done by paying attention to whether the individual performs the specified function on time, receives help or needs an assistive device. If the desired function is performed completely with help, 1 point is given; if the individual performs it completely independently, safely and at the appropriate time, 7 points are given. Accordingly, the individual receives at least 18 points, which means that he/she is fully dependent. The maximum full score that can be obtained from the scale is 126, which means that the individual is fully independent.
Modified Ashworth Scale (MAS) | First day
  The 'Modified Ashworth Scale (MAS)' scores spasticity on a scale ranging from "0" to "4" according to the definition of velocity-dependent spasticity. High MAS score indicates severe spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Keklikci, Res. Assist., Principal Investigator — Alanya Alaaddin Keykubat University
Locations (1):
- Alanya Alaaddin Keykubat University, Antalya, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No